CLINICAL TRIAL: NCT06890039
Title: Phase II, Double-blind, Randomized, Placebo-controlled, Multicentre Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of TAK-242 and (G-CSF) in Subjects With (sAH) and (ACLF)
Brief Title: A-TANGO Phase 2 Study
Acronym: A-TANGO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yaqrit Ltd (Industry)
Collaborators: European Foundation for Study of Chronic Liver Failure (Other); University College, London (Other); HEPYX LIMITED (Unknown); CROWDHELIX LIMITED (Unknown); Charite University, Berlin, Germany (Other); University of Leipzig (Other); Concentris research management gmbh (Unknown); Assistance Publique - Hôpitaux de Paris (Other); Leiden University Medical Center (Other); INTERNATIONAL MARKET ACCESS CONSULTING GMBH (Unknown); KlinEra Global Services (Industry); European Association for the Study of the Liver (Unknown); EUROPEAN LIVER PATIENTS' ASSOCIATION (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G-TAK-ES-01; 945096 (Other Grant/Funding Number: EUROPEAN COMMISSION H2020); 2022-000128-39 (EudraCT Number); 1005490 (Other: IRAS)
Record Dates: First submitted 2024-12-13; First posted 2025-03-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute-On-Chronic Liver Failure; Alcoholic Hepatitis; Liver Cirrhosis, Alcoholic
Keywords: Novel combinatorial therapy; Improve hepatocyte proliferation; ACLF; Liver disease
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis, Alcoholic; Liver Cirrhosis, Alcoholic; Liver Diseases | interventions — ethyl 6-(N-(2-chloro-4-fluorophenyl)sulfamoyl)cyclohex-1-ene-1-carboxylate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: This study is randomized, double-blind, and placebo-controlled to avoid subjective bias in the assessment of the study drug. Placebo will be administered as a control in order to establish the frequency or magnitude of changes in clinical endpoints that may occur with standard supportive care, in the absence of active experimental treatment.
Who Masked: Participant, Investigator
Masking Description: The investigational drug blind is maintained by study drug/placebo preparation by an unblinded person (hospital pharmacist, or equivalent).
  The study drug blind shall not be broken by the investigator unless information concerning the study drug is necessary for the medical treatment of the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care (SOC) plus placebo for TAK-242 plus placebo for G-CSF (Placebo Comparator)
  Interventions: Drug: Placebo
- Standard of care (SOC) plus TAK-242 plus placebo for G-CSF (Active Comparator)
  Interventions: Drug: TAK-242
- Standard of Care (SOC) plus TAK-242 plus G-CSF (Active Comparator)
  Interventions: Drug: TAK-242; Drug: G-CSF (Filgrastim)

INTERVENTIONS:
Drug: Placebo — Matching placebo for TAK-242: 5% dextrose solution and commercially available 20% intralipid (prepared by hospital pharmacy staff)
  Matching placebo for G-CSF: identical to vehicle for filgrastim (prepared for injection by hospital pharmacy staff)
  Arms: Standard of care (SOC) plus placebo for TAK-242 plus placebo for G-CSF
Drug: TAK-242 — TAK-242 concentrate for solution for infusion (80 mg/ mL in 3 mL ethanol) ): 240 mg TAK-242 per vial. To be reconstituted with 5% dextrose (36 mL) and commercially available 20% intralipid (21 mL).
  TAK-242) will be administered as a continuous IV infusion starting with a loading dose of 0.9 mg/kg administered over 30 minutes, followed by a continuous, constant rate infusion of 1.8 mg/kg/day for 10 days.
  PLUS placebo for G- CSF
  Arms: Standard of Care (SOC) plus TAK-242 plus G-CSF; Standard of care (SOC) plus TAK-242 plus placebo for G-CSF
Drug: G-CSF (Filgrastim) — Commercially available vials for subcutaneous injection. Quantitative composition (per mL):
  Filgrastim: 300 mcg Acetate: 0.59 mg Sorbitol: 50.0 mg Tween® 80: 0.04 mg Sodium: 0.035 mg Water for Injection USP q.s. ad 1.0 mL
  G-CSF will be given subcutaneously once daily at a dose of 5 µg/kg for 5 days (Day 1-5) and at Day 8 (6 injections in total)
  Arms: Standard of Care (SOC) plus TAK-242 plus G-CSF

SUMMARY:
The purpose of this research is to know if a new combination of drugs (TAK-242 and G-CSF) in combination with standard therapy for acute-on-chronic liver failure (ACLF) is more effective than standard therapy for ACLF treatment and is safe.

Description of the population to be studied: ACLF is a syndrome that occurs in patients with chronic liver disease, with or without previously diagnosed cirrhosis, which is characterized by acute hepatic decompensation. Cirrhosis is a chronic disease of the liver marked by degeneration of cells, inflammation, and thickening and scarring (fibrosis) of liver tissue. Hepatic decompensation is a sudden decline in liver function. It is characterized by severe liver damage and complications like jaundice (yellowing of the skin or whites of the eyes), ascites (a condition where excess fluid accumulates in the abdominal cavity and in abdominal organs) and encephalopathy (a group of symptoms that result from damage or dysfunction in the brain, causing a range of cognitive and neurological impairments). It may result in liver failure, one or more organ failures other than liver (renal, brain, coagulation, respiratory, cardiovascular), and is associated with increased mortality within 28-days and up to 3 months from onset. Grade 1 ACLF has a >15% risk of mortality at 28 days.

Purpose of the study: The investigational medication, TAK-242, is aimed at stopping an "over-reaction" of the immune system (the body's defense system) while G-CSF encourages your liver cells to grow. In patients with severe inflammation of the liver due to alcohol [severe alcoholic hepatitis (sAH)] and ACLF, this over-reaction may cause the liver and other organs in the body to suddenly stop working (organ failure). The hypothesis of the study is that by blocking this over-reaction and encouraging your liver cells to grow your condition may improve.

DETAILED DESCRIPTION:
The purpose of this Phase 2 clinical trial is to investigate

* the safety of TAK-242 alone or in combination with G-CSF (G-TAK) in patients with sAH and ACLF.
* the effect of TAK-242 alone or in combination with G-CSF (G-TAK) on the disease severity of ACLF.

Study design:

Multi-center, randomized, double-blind, placebo-controlled trial. Study drug will be administered while subjects are hospitalized. Patients will have been hospitalized for their underlying disease.

78 patients to be randomized (1:1:1) to one of the following three arms:

* Standard of care (SOC) plus placebo for TAK-242 plus placebo for G-CSF
* Standard of care (SOC) plus continuous IV infusion of TAK-242 for 10 days (Day 1-10) plus placebo for G-CSF.
* Standard of Care (SOC) plus continuous IV infusion of TAK-242 for 10 days (Day 1-10) plus daily subcutaneous G-CSF injections for 5 days (Day 1-5) and at Day 8 (6 injections in total)

Follow-up visits will occur on Day 14 (± 4 d), Day 28 (± 5 d), and Day 84 (± 7d). For each patient, the total duration of subject participation in the study, including screening, will be 86 ± 7 days.

The total study duration is estimated to be approximately 42 months from screening of first patient until study completion of the last patient/last visit and data analysis.

The placebo is the same as the investigational medication but does not contain the active ingredient. A placebo is used to check that any effects seen in people taking part in the study are because of the investigational medications and not due to the underlying disease (for safety) or to spontaneous improvement (for efficacy)

The study will also look at how the investigational medications affect the body (known as "pharmacodynamics") and how your body processes the investigational medications (known as "pharmacokinetics").

Investigational product:

* TAK-242 concentrate for solution for infusion (80 mg/mL in 3 mL ethanol): 240 mg TAK-242 per vial. To be reconstituted with 5% dextrose (36 mL) and commercially available 20% intralipid (21 mL).
* Matching placebo: 5% dextrose solution and commercially available lipid emulsion (prepared in hospital pharmacy
* G-CSF(filgrastim): Commercially available vials for subcutaneous injection. Matching placebo: identical to vehicle for filgrastim (prepared for injection by hospital pharmacist, or equivalent)

Management of patients Management of patients enrolled in the study will be performed according to guidelines and best practice of treatments for the management of complications of cirrhosis derived from international societies. Standard medical therapy also means that patients will be clinically assessed daily, including results of clinical chemistry and blood count.

An independent Data and Safety Monitoring Board (DSMB)will review safety and pharmacokinetic data after randomization of 18 patients (n=6 in each treatment arm) with complete PK analysis through Day 4 (±1 d). The DSMB will assess the relevance of drug-related adverse events and drug-drug interactions.

Compliance with Good Clinical Practices The study will be conducted in accordance with all applicable aspects of GCP. Statistical Analysis of Data The primary endpoint - safety - will be evaluated by descriptive statistics.

Secondary endpoints will offer an indication about potential signals in efficacy for future trials. Sample size was estimated to find differences in CLIF-C OF score between G-TAK and placebo, to allow a 90% statistical power to detect a 1.5-point difference between the combination G-TAK and the SOC arm in the reduction of CLIF-C OF score after 14 days from trial enrolment. A 5% Type-I error for a two-sided Student's t-test with repeated measurements is assumed. This sample size includes a dropout rate of 15%.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for inclusion into the study must meet all of the following criteria:

  1. Male and female subjects ≥18 of age and ≤75 years of age
  2. Compliance with acceptable contraceptive methods.
  3. With a diagnosis of severe alcoholic hepatitis that is resistant to steroid therapy as defined by a Lille score of >0.45 and/or in whom steroids are contraindicated.
  4. Eligible subjects will have Grade 1-3 ACLF with a maximum of three organ failures using the CLIF-C OF score AND the CLIF-C ACLF-CRP score of >35 and <60.

Exclusion Criteria:

* Patients with any of the following criteria are to be excluded:

  * Refusal to give informed consent
  * Mechanical ventilation due to respiratory failure and/or need for renal replacement therapy and or requiring inotropes for circulatory support with a noradrenaline requirement of >0.5ug/kg/min to maintain mean arterial pressure > 70mmHg
  * Subject has received any investigational drug within 30 days of randomization
  * Subject has any of the following conditions:

    * history of liver transplantation
    * postoperative decompensation after partial hepatectomy
    * liver failure without underlying chronic liver injury
  * Any untreated infections (<48h antibiotic therapy) including gram-positive infections, active tuberculosis or coinfection with HIV.
  * Chronic or pre-existing kidney failure, survival prognosis of <6 months due to severe co-morbid conditions that might confound study results or compromise subject safety
  * Methemoglobinemia, clinically-significant disseminated intravascular coagulation, uncontrolled bleeding, sickle cell anemia
  * Uncontrolled seizures, Creutzfeldt-Jakob disease, glucose-6-phosphate dehydrogenase deficiency.
  * Active malignancy, premalignant hematological disorders (e.g., myelodysplastic syndrome, chronic myeloid leukemia) or multiorgan failure (≥ 4 organ failures).
  * Pregnancy or nursing women
  * Allergy to eggs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of TAK-242 in combination with G-CSF and alone in subjects with sAH and ACLF compared to placebo | Baseline to Day 14
  To assess the safety of TAK-242 in combination with G-CSF (G-TAK) and alone in subjects with sAH and ACLF compared to placebo from baseline to Day 14:
  * The percentage of subjects who experience at least 1 treatment-emergent AE (TEAE) or SAE.
  * The percentage of subjects who discontinue the study drug due to an AE (including methemoglobinemia).

SECONDARY OUTCOMES:
Changes in CLIF-C OF score | Baseline to Day 14
  Changes in CLIF-C OF score in subjects treated with G-TAK compared with placebo from baseline to Day 14 CLIF-C OF (Chronic Liver Failure Organ Failure) - The CLIF-C organ failure (OF) score is used to diagnose acute-on-chronic liver failure (ACLF) in patients with acute decompensation of cirrhosis. Each organ system is scored on a scale to generate the overall CLIF-C OF score, ranging from 0 to 18. A higher CLIF-C OF score translates into a higher ACLF grade.
Changes in CLIF C ACLF-CRP score | Baseline to Day 84
  Changes in CLIF-C OF score in patients treated with TAK-242 alone compared with G-TAK and placebo, as well as changes in CLIF C ACLF-CRP score between all arms
  CLIF-C Acute-on-chronic liver failure - c-reactive protein (CLIF-C ACLF-CRP) will be calculated using this formula:
  CLIF-C ACLF-CRP score = 10 x (0.293 x CLIF-C OF score + 0.034 x Age[years] + 0.292 x log(CRP) - 0.8)
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  tmax(hr): Time point where the peak plasma concentration is maximum will be calculated
To Investigate the effects of TAK-242 alone or in combination with G-CSF, compared with placebo and between active treatment groups, on key biomarkers for inflammation, cell death, liver function, regeneration and senescence | From Baseline to Day 4, 7, and 14
  Changes from baseline after 14 days in naturally log-transformed key liver function biomarkers will include:
  * total bilirubin (TB)
  * cleaved Cytokeratin-18 (M30)/ Cytokeratin-18 (M65)
  * transforming growth factor beta 1 (TGFb1)
  * interleukin 22 (IL-22)
  * interleukin 22 binding protein (IL-22BP)
  * C-reactive protein (CRP)
  * hepatic growth factor (HGF)
  * stromal cell-derived factor 1 (SDF-1),
  * soluble urokinase-type plasminogen activator receptor (suPAR))
  * DNA methylation
  * circulating RNAs (genes MYLK3, SLC22A13, TPRG1-AS1, AC020633.1, TPRG1-AS1, NUDT4P1 Biomarkers of Humoral Inflammation and Cell Death, Cellular inflammation, regeneration & senescence, metabolic and genetics and mitochondrial function are assessed individually between treatment groups as well as overall, global trends between treatment groups. They are not aggregated to arrive at one reported value.
To investigate transplant free and overall survival in subjects with sAH and ACLF | Upto Day 84
  To investigate the effect of TAK-242 alone or the combination of TAK-242 and G-CSF (G-TAK) versus placebo on Day 28 and Day 84 transplant free and overall survival in subjects with sAH and ACLF.
  This is not a scale. Patients either do or do not have a liver transplant during the study period; and either survive or don't survive.
Change in organ function between different treatment arms. | Baseline to Day 14
  Assessments of organ failure, systemic inflammation, and ACLF
To investigate the effect on the Quality of Life | Baseline to Day 84
  To investigate the effect of TAK-242 alone or the combination G-TAK compared with placebo and each other on the Quality of Life in subjects with sAH and ACLF. The scoring system that will be used is EQ5D5L, which allows assessment of QoL changes in sick patients
  Quality of Life scale is scored from 0 to 100, with 0 being worst health you can imagine; 100 best health.
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  t1/2(hr) will be determined from the terminal phase in plasma after drug administration
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  Cmax(ng/mL): highest concentration of a drug in the blood will be calculated
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  Steady-state concentration (Cssng/mL) will be calculated for drug being absorbed in the body when the drug is given continuously or repeatedly
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  AUC last (h*ng/ml): Area under curve from pre-dose to the last sampling time-point will be calculated
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  AUC infinity (h*ng/ml): Area under curve from pre-dose to the extrapolated data till the concentration reaches to baseline
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  Total body clearance (L/h) will be calculated
Pharmacokinetics parameters for TAK-242 along with its two main metabolites and G-CSF | Baseline to Day 7
  Total body clearance at steady state (L/h) will be calculated